CLINICAL TRIAL: NCT02414568
Title: A Prospective Phase II Study of Bendamustine in Patients Aged Over 60 Years With Classical Hodgkin Lymphoma Treated by Prednisone, Vinblastine and Doxorubicin
Brief Title: Bendamustine Study in Classical Hodgkin Lymphoma Patients Over 60 Treated by Prednisone, Vinblastine and Doxorubicin
Acronym: PVAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVAB
Record Dates: First submitted 2015-03-30; First posted 2015-04-10 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — Bendamustine Hydrochloride; Prednisone; Vinblastine; Doxorubicin

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVAB regimen (Experimental): Prednisone 40 mg/m2 (PO) Days 1-5 ; Vinblastine 6 mg/m2 (IV) Day 1 ; Doxorubicin 40 mg/m2 (IV) Day 1 ; Bendamustine 120 mg/m2 (IV) Day 1
  Interventions: Drug: Bendamustine; Drug: Prednisone; Drug: Vinblastine; Drug: Doxorubicin

INTERVENTIONS:
Drug: Bendamustine — Bendamustine 120 mg/m2 (IV) Day 1
  Other Names: LEVACT
Drug: Prednisone — Prednisone 40 mg/m² PO
  Other Names: CORTANCYL
Drug: Vinblastine — Vinblastine 6 mg/m² IV
  Other Names: VELBE
Drug: Doxorubicin — Doxorubicin 40 mg/m² IV
  Other Names: ADRIBLASTINE

SUMMARY:
This study evaluates bendamustine in patients aged over 60 years with classical Hodgkin Lymphoma treated by prednisone, vinblastine and doxorubicin. 90 patients will be enrolled in this study.

DETAILED DESCRIPTION:
The usual treatment for Hodgkin lymphoma is chemotherapy Adriamycin (also known as doxorubicin) + Bleomycin + Vinblastine + Dacarbazine (ABVD). Studies have shown that patients aged over 60 years have a lower tolerance and efficiency during this treatment than younger patients. There are particular pulmonary toxicities with bleomycin included in the ABVD treatment.

Alternative treatment strategies have been proposed removing bleomycin in the Prednisone + Vinblastine + Adriamycin/Doxorubicin +Gemcitabine (PVAG) protocol evaluated in more than 60 patients. Compared to ABVD treatment, PVAG treatment presented a more favorable toxicity profile. The quality of response between the two treatments is substantially equal.

Bendamustine was evaluated in four studies in patients with Hodgkin lymphoma in relapse and showed higher efficacy than gemcitabine with an acceptable toxicity profile.

In this study, the Sponsor and the coordinating investigator propose to replace dacarbazine in the standard ABVD protocol by bendamustine and to stop using bleomycin.

The main objective of this study is to evaluate the safety and efficacy of bendamustine in patients treated with prednisone, vinblastine and doxorubicin. This is the PVAB treatment with which LYSARC and the coordinating investigator expect better tolerability and quality response.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a first diagnosis of classical Hodgkin lymphoma according to the World Health Organization (WHO) criteria excluding nodular lymphocyte predominant subtype
* Age of 61 years or older
* No previous treatment for Hodgkin lymphoma
* Ann Arbor stages:

  * II with mediastinum/thorax ≥0.33 or extranodal localization and with B symptoms
  * Or III
  * Or IV
* Baseline 18-FluoroDeoxyGlucose (FDG) PET scan (PET0) performed before any treatment with at least one hypermetabolic lesion
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate cardio-pulmonary function with Left Ventricular Ejection Fraction (LVEF) ≥ 50%
* Adequate renal function with creatinine clearance ≥ 40 mL/mn (MDRD formula)
* For patients aged 70 years old and more, a Mini Nutritional Assessment (MNA) ≥ 17
* A minimum life expectancy of 3 months
* Negative Human Immunodeficiency Virus, Hepatitis B (HB) Virus (anti-HB c negativity) and Hepatitis C Virus serologies tests ≤ 30 days before inclusion (except after vaccination)
* Having previously signed a written informed consent
* The patient must be covered by a social security system, if applicable
* Men patient must agree to use an adequate method of contraception during the study treatment and until 6 months after the end of the study treatment.

Exclusion Criteria:

* Any other type of lymphoma including nodular lymphocyte predominant subtype
* Any history of treated Hodgkin lymphoma
* Contra-indication to any drug contained in the chemotherapy regimens
* Any serious active disease (according to the investigator's decision)
* Poor hepatic function (total bilirubin level > 30 μmol/L or transaminases > 2.5 maximum normal level) unless these abnormalities are related to the lymphoma
* Poor bone marrow reserve as defined by leukocytes < 2 G/L or platelets < 100 G/L, unless related to bone marrow infiltration
* Any history of cancer during the last 3 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma. Patients previously diagnosed with prostate cancer are eligible if they fulfil all the followings:

  1. their disease was T1-T2a, N0, M0, with a Gleason score ≤ 7, and a prostate specific antigen (PSA) ≤ 10 ng/mL prior to initial therapy,
  2. they had definitive curative therapy (i.e. prostatectomy or radiotherapy) ≥ 2 years before Day 1 of Cycle 1,
  3. at a minimum 2 years following therapy, they had no clinical evidence of prostate cancer and their PSA was undetectable if they underwent prostatectomy or < 1 ng/mL if they did not undergo prostatectomy
* Severe metabolic disease interfering with normal application of protocol treatment as uncontrolled diabetes mellitus leading to impossibility to perform PET scan
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study
* Adult under tutelage

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Complete Metabolic Response rate at the end of study treatment (after 6 cycles of study treatment or at premature treatment discontinuation) defined according to Lugano Classification | 3 years
  Complete Metabolic Response rate at the end of study treatment (after 6 cycles of study treatment or at premature treatment discontinuation) defined according to Lugano Classification

SECONDARY OUTCOMES:
Feasibility of the protocol, with adequate protocol adherence (adequate dose without excessive delay) | 5 years
  Feasibility of the protocol, with adequate protocol adherence (adequate dose without excessive delay)
Safety profile including immediate toxicities and non-tumor events | 5 years
  Safety profile including immediate toxicities and non-tumor events
Progression-free survival | 5 years
  Progression-free survival
Disease-free survival | 5 years
  Disease-free survival
Overall survival | 5 years
  Overall survival
Geriatric assessment program | 5 years
  7 Quality of Life Questionnaires (QLQ)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Ghesquières, MD, Principal Investigator — The Lymphoma Academic Research Organisation
Locations (40):
- Belgium (4):
  - A. Z. Sint-Jan, Bruges
  - Clinique Universitaire St Luc, Brussels
  - CHU de Liège, Liège
  - UCL Mont Godinne, Yvoir
- France (36):
  - CHU d'Amiens - Groupe Hospitalier Sud, Amiens
  - Hôpital Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHRU de Brest - Hôpital Morvan, Brest
  - CHU de Caen, Caen
  - Médipôle de Savoie, Challes-les-Eaux
  - CH Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU Dijon - Hôpital d'Enfants, Dijon
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CH Départemental Vendée, La Roche-sur-Yon
  - CH de Versailles, Le Chesnay
  - CH du Mans, Le Mans
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CHR de Metz-Thionville - Hôpital de Mercy, Metz
  - Hôpital Lapeyronie, Montpellier
  - CH de Mulhouse, Mulhouse
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHRU de Nîmes, Nîmes
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Necker, Paris
  - CHU de Bordeaux - Hôpital Haut Lévêque - Centre François Magendie, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - CH Rene Dubos, Pontoise
  - Centre Hospitalier Annecy-Genevois - Site d'Annecy, Pringy
  - CHU de Reims, Reims
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Tours - Hôpital Bretonneau, Tours
  - CH de Valenciennes, Valenciennes
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghesquieres H, Krzisch D, Nicolas-Virelizier E, Kanoun S, Gac AC, Guidez S, Touati M, Laribi K, Morschhauser F, Bonnet C, Waultier-Rascalou A, Orsini-Piocelle F, Andre M, Fournier M, Morand F, Berriolo-Riedinger A, Burroni B, Damotte D, Traverse-Glehen A, Quittet P, Casasnovas O. The phase 2 LYSA study of prednisone, vinblastine, doxorubicin, and bendamustine for untreated Hodgkin lymphoma in older patients. Blood. 2024 Mar 14;143(11):983-995. doi: 10.1182/blood.2023021564. PMID 37979133